CLINICAL TRIAL: NCT06871228
Title: DIscontinuation of Anticoagulation With Intensive Rhythm MONitoring CompareD With Continuous Anticoagulation in Post-ablation Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Discontinuation of Anticoagulation With Intensive Rhythm Monitoring in Post-ablation Patients With Atrial Fibrillation
Acronym: DIAMOND-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KLS09
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; catheter ablation; smartwatch; anticoagulation; thromboembolism; bleeding
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of NOACs (Experimental): Participants randomized to the experimental arm will stop oral anticoagulation (NOACs) immediately after randomization. All participants in this trial (including this arm) will undergo intensified rhythm surveillance using a smartwatch capable of single-lead ECG plus scheduled Holter or single-lead ECG patch monitoring (at least every 6 months; every 2 months encouraged), with symptom-triggered and opportunistic ECGs. AF recurrence is defined as ECG-documented AF/AFL/atrial tachycardia lasting ≥30 seconds.
  Interventions: Drug: NOAC discontinuation; Device: Smartwatch single-lead ECG monitoring
- Continuation of NOACs (Active Comparator): Participants randomized to the control arm will continue NOAC therapy after randomization. The same intensified rhythm monitoring approach (smartwatch ECG plus scheduled Holter/patch and symptom/opportunistic ECG confirmation) applies.
  Interventions: Drug: NOAC continuation; Device: Smartwatch single-lead ECG monitoring

INTERVENTIONS:
Drug: NOAC discontinuation — Stop NOACs immediately after randomization (experimental arm)
  Arms: Discontinuation of NOACs
Drug: NOAC continuation — Continue guideline-recommended NOAC therapy after randomization (control arm)
  Arms: Continuation of NOACs
Device: Smartwatch single-lead ECG monitoring — Continuous AF screening with a smartwatch capable of recording single-lead ECG, with ECG confirmation required for diagnosis (PPG abnormalities alone are not diagnostic).

SUMMARY:
DIAMOND-AF is a multicenter, randomized, open-label trial evaluating whether discontinuing oral anticoagulation after successful atrial fibrillation ablation can reduce bleeding risk without increasing death or thromboembolism risks. Adults aged 18-80 years, 60-365 days post-ablation, with CHA2DS2-VA ≥2, no prior stroke/TIA/systemic embolism, continuous NOAC use, and no documented atrial tachyarrhythmia recurrence will be randomized 1:1 to stop NOACs immediately or to continue NOAC therapy. All participants use intensified rhythm surveillance including smartwatch ECG and Holter/patch monitoring (at least every 6 months; every 2 months encouraged) to detect recurrence. Co-primary endpoints are (1) non-inferiority for the composite of all-cause death, ischemic stroke, or systemic embolism and (2) superiority for the composite of ISTH major bleeding or ISTH clinically relevant non-major bleeding. The planned sample size is 4,100 participants.

DETAILED DESCRIPTION:
DIAMOND-AF is an investigator-initiated, multicenter, randomized, open-label, parallel-group trial designed to evaluate post-catheter ablation anticoagulation management in patients with atrial fibrillation (AF/AFL). The trial will enroll adults aged 18-80 years who are 60±15 to 365±15 days after AF ablation, have a CHA2DS2-VA score ≥2, have no history of ischemic stroke/transient ischemic attack/systemic embolism, have been continuously taking a non-vitamin K antagonist oral anticoagulant (NOAC), and have no documented atrial tachyarrhythmia recurrence after ablation. Eligible participants will be randomized 1:1 to (1) discontinue NOAC immediately after randomization or (2) continue NOAC therapy. The study uses a co-primary endpoint strategy: a non-inferiority assessment for the composite efficacy endpoint (all-cause death, ischemic stroke, or systemic embolism) and a superiority assessment for the composite safety endpoint (ISTH major bleeding or ISTH clinically relevant non-major bleeding). To maximize safety while testing an anticoagulation-discontinuation strategy, all participants will undergo intensified rhythm monitoring using a smartwatch capable of single-lead ECG plus scheduled Holter/single-lead ECG patch monitoring (at least every 6 months; every 2 months encouraged), with symptom-triggered and opportunistic ECGs incorporated. AF Recurrence is defined as any ECG-confirmed atrial tachyarrhythmia (AF/AFL/atrial tachycardia) lasting ≥30 seconds; once AF recurrence is confirmed, the participant will be censored and will exit further trial follow-up. Participants will have in-person/structured study visits at months 3 and 6 after randomization, then every 6 months, with additional rhythm/anticoagulation follow-up every 2 months. The planned sample size is 4,100 participants (2,050 per group).

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

1. Age 18 to 80 years.
2. 60±15 to 365±15 days after atrial fibrillation/atrial flutter (AF/AFL) ablation.
3. CHA2DS2-VA score ≥2.
4. No history of stroke, transient ischemic attack (TIA), or systemic embolism.
5. Continuous use of a NOAC since AF/AFL ablation.
6. No documented atrial tachyarrhythmia recurrence since ablation.
7. No antiarrhythmic drug (AAD) use within the past 2 months.
8. Able and willing to provide written informed consent.
9. Able and willing to comply with study procedures and follow-up.

Exclusion Criteria

Participants will be excluded if any of the following criteria are present:

1. High risk of post-ablation recurrence (e.g. including premature atrial contraction burden >3% on any ambulatory ECG/Holter recording).
2. Moderate-to-severe mitral stenosis (mitral valve area ≤2.0 cm²) or mechanical heart valve.
3. Increased bleeding risk, including any of the following:

   1. Current ISTH major bleeding or clinically relevant non-major bleeding (CRNMB).
   2. History of non-traumatic major bleeding (e.g., intracranial, intraocular, spinal, retroperitoneal, gastrointestinal, or intra-articular) unless the reversible cause has been permanently eliminated.
   3. Unresolved intracranial aneurysm/vascular malformation, or active/unhealed gastric or duodenal ulcer.
   4. General anesthesia surgery within the past 3 months.
   5. Planned surgery within the next 3 months.
   6. Known bleeding diathesis (e.g., hemophilia).
   7. Uncontrolled hypertension (SBP >180 mmHg and/or DBP >110 mmHg).
   8. Hemoglobin <90 g/L or blood transfusion within 4 weeks prior to enrollment.
   9. Platelet count <50 × 10⁹/L.
   10. End-stage kidney disease (eGFR <15 mL/min/1.73 m²) or on dialysis.
   11. Severe liver disease (e.g., esophageal variceal bleeding, ascites, hepatic encephalopathy, or jaundice).
   12. Known intolerance to oral anticoagulants or contraindication to oral anticoagulation.
4. Any condition requiring continued oral anticoagulation (e.g., pulmonary embolism, deep vein thrombosis, hypertrophic cardiomyopathy, cardiac amyloidosis).
5. Conditions associated with high non-cardioembolic stroke risk, including carotid, vertebral, or intracranial arterial stenosis ≥70%.
6. Prior left atrial appendage (LAA) occlusion, surgical LAA excision/closure, or intraoperative confirmation of LAA electrical isolation.
7. Female participants who are pregnant or breastfeeding, or of childbearing potential not using effective contraception.
8. Life expectancy <2 years.
9. Current participation in another interventional clinical trial.
10. Any condition that, in the investigator's judgment, would make the participant unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4100 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of all-cause death, ischemic stroke, or systemic embolism | 48 months
  The primary effectiveness outcome is to determine whether NOAC discontinuation with intensified rhythm monitoring is non-inferior to continued NOAC therapy for the composite of all-cause death, ischemic stroke, or systematic embolism.
  Ischemic stroke is defined as an acute focal dysfunction from CNS infarction lasting ≥24h, with potential hemorrhagic transformation. Systemic embolism refers to arterial embolism or thrombosis (excluding stroke or TIA).
ISTH major bleeding or ISTH clinically relevant non-major bleeding | 48 months
  The primary safety outcome is to determine whether NOAC discontinuation is superior to continued NOAC therapy in reducing the composite of ISTH major bleeding or ISTH clinically relevant non-major bleeding (CRNMB).
  ISTH major bleeding and CRNMB are defined per ISTH criteria (e.g., fatal bleeding; critical-site bleeding; hemoglobin drop ≥20 g/L or transfusion ≥2 units for major bleeding; and medically attended, hospitalization-escalating, or unplanned-visit bleeding for CRNMB).

SECONDARY OUTCOMES:
All-cause death | 48 months
Ischemic stroke | 48 months
Systemic embolism | 48 months
Major bleeding | 48 months
Clinically relevant non-major bleeding | 48 months
  Clinically relevant non-major bleeding is defined as any sign or symptom of hemorrhage that does not meet the criteria for the ISTH definition of major bleeding, but meets at least one of the following criteria:
  1. Requiring medical intervention by a healthcare professional.
  2. Leading to hospitalization or increased level of care.
  3. Prompting a face-to-face evaluation by a healthcare provider.
Cardiovascular death | 48 months
Atrial Fibrillation Effect on Quality-of-Life questionnaire (AFEQT) score | 48 months
  The AFEQT score ranges from 0 to 100, with higher scores indicating better QoL.
Atrial fibrillation Recurrence | 48 months
  Defined as atrial tachyarrhythmia lasting ≥30s on ECG
Five-Level EuroQol Five Dimensions Questionnaire (EQ-5D-5L) score | 48 months
  The EQ-5D-5L measures health-related quality of life. It has two parts: 1) a 5-dimension descriptive system (mobility, self-care, usual activities, pain, anxiety/depression) with 5 levels per dimension, generating a utility value; 2) a Visual Analogue Scale (VAS) from 0 (worst) to 100 (best) for overall health. Higher scores indicate better health.
Generalized Anxiety Disorder-7 item questionnaire (GAD-7) score | 48 months
  Anxiety is measured by GAD-7 score, with scores ranging from 0 to 21, where higher scores indicate greater levels of anxiety.
Patient Health Questionnaire-9 item questionnaire (PHQ-9) score | 48 months
  Depression is evaluated using PHQ-9 score, which is scored from 0 to 27, with a higher score indicating greater levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, MD, Principal Investigator — Beijing Anzhen Hospital; Caihua Sang, Principal Investigator — Beijing Anzhen Hospital
Locations (19):
- China (19):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Luohe Central Hospital, Luohe, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Liaocheng Heart Hospital, Liaocheng, Shandong
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No